CLINICAL TRIAL: NCT05124548
Title: Sleep Characteristics in Post-Corona Virus Disease 2019 Patients Compared to Healthy Controls - An Observational Trial
Brief Title: Sleep Characteristics in Post-COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Rembert Koczulla, Principal investigator, Schön Klinik Berchtesgadener Land
Other Study IDs: WHOOP Sleep
Record Dates: First submitted 2021-11-17; First posted 2021-11-18 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Post-COVID-19
Keywords: SARS-CoV-2 infection; REM sleep; Chronic fatigue; Whoop strap; Polysomnography
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-COVID condition
  Interventions: Diagnostic Test: Sleep diagnostics
- Healthy controls
  Interventions: Diagnostic Test: Sleep diagnostics

INTERVENTIONS:
Diagnostic Test: Sleep diagnostics — On study day 4, all participants perform a single night sleep assessment in a sleep lab via Polysomnography (PSG) and WHOOP strap, a digital Fitness and health Coach.

SUMMARY:
After acute infection, patients with coronavirus disease 2019 (COVID-19) often suffer from persisting symptoms for more than 3 months (post COVID-19). Sleep disorders (31%) have already been assessed by questionnaires and interviews in post-COVID-19, but have not yet been proven by polysomnography (PSG), the gold standard for sleep testing. This study aimed to measure sleep characteristics in post-COVID-19 patients.

DETAILED DESCRIPTION:
Hypothesis: We hypothesize that post-COVID-19 patients have a significantly higher apnea-hypopnea index (AHI) during sleep compared to healthy controls.

15 post-COVID-19 patients and 15 healthy controls will perform a baseline assessment on day 1 including a 1-minute sit-to-stand test (STST), post-COVID functional scale (PCFS), Ordinal Scale for Clinical Improvement (OSCI), history of COVID-19, social anamnesis, Pittsburgh Sleep Questionnaire and subjective limitations of sleep.

On day 4, after an initialization phase for WHOOP strap (a digital fitness and health coach), all patients performed a single night sleep assessment in a sleep lab via Polysomnography and WHOOP.

ELIGIBILITY:
Inclusion Criteria:

Post-COVID-19 Group:

* Patients after SARS-CoV-2 infection with signs of Post-COVID-19
* ≥18 years
* written informed consent

Healthy controls:

* No history of SARS-CoV-2 infection
* ≥18 years
* written informed consent

Exclusion Criteria:

Post-COVID-19 Group:

* Diagnosis of a breathing-related sleep disorder before SARS-CoV-2 infection
* BMI >25kg/m2

Healthy controls:

* Diagnosis of a breathing-related sleep disorder
* BMI >25kg/m2

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: 30 patients will be included in this study. Patients with Post-COVID-19 (n=15) are characterized by Symptoms usually starting 3 months following the onset of COVID-19 that last for at least 2 months and cannot be explained by an alternative diagnosis than SARS-CoV-2 infection.
  Healthy controls are characterized by having no history of SARS-CoV-2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea-Index (AHI) | One single night on study day 4
  Number of apnea or hypopnea Events per hour of sleep

SECONDARY OUTCOMES:
Rapid Eye Movement (REM) sleep phase | One single night on study day 4
  Duration of REM sleep Phase (minutes)
Deep sleep phase | One single night on study day 4
  Duration of deep sleep Phase (minutes)
Light sleep phase | One single night on study day 4
  Duration of light sleep Phase (minutes)
Periodic leg movement Index | One single night on study day 4
  Number of Periodic leg movements per hour of sleep
Obstructive apnea | One single night on study day 4
  Number of obstructive apnea Events per night
Central apnea | One single night on study day 4
  Number of central apnea Events per night
Mixed apnea | One single night on study day 4
  Number of mixed apnea Events per night

CONTACTS AND LOCATIONS:
Locations (1):
- Schoen Klinik Berchtesgadener Land, Schönau am Königssee, Germany